CLINICAL TRIAL: NCT02355548
Title: Rapid Risk Stratification for Outpatient Treatment of Low-risk Pulmonary Embolism
Brief Title: Outpatient Treatment of Low-risk Pulmonary Embolism
Acronym: Low Risk PE
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1018558
Record Dates: First submitted 2014-11-18; First posted 2015-02-04 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Outpatient Treatment: All patients eligible for the study will have their PE treated in the outpatient setting.
  Interventions: Other: Outpatient Treatment of Pulmonary Embolism

INTERVENTIONS:
Other: Outpatient Treatment of Pulmonary Embolism — Patients who participate in the study will be treated for their pulmonary embolism in an outpatient setting instead of being hospitalized.

SUMMARY:
This study is looking at the safety and effectiveness of treating Patients diagnosed with a low-risk Pulmonary Embolism (PE) in an outpatient setting instead of the standard, in-patient hospitalization. Patients have several medical tests done during their Emergency Department visit. Based on those tests, those who are determined to have a low-risk PE are eligible to participate in the study. Those choosing to participate are discharged after 12 hours of medical observation. Patients who choose to participate are followed up by telephone approximately 90 days later.

ELIGIBILITY:
Inclusion Criteria:

1. Pulmonary Embolism, diagnosed by CTA or high probability VQ Scan
2. Total Pulmonary Embolism Severity Index (PESI) score <86

Exclusion Criteria:

1. Massive Pulmonary Embolism: Hypotension with signs of right heart strain on CTA or Echocardiogram
2. Sustained Systolic Blood Pressure (SBP) <95 mmHg during Emergency Department or observation stay.
3. Age <18
4. Pregnant
5. Renal insufficiency (Creatinine Clearance <30)
6. Hepatic Dysfunction (AST/ALT/ALP > 3 times upper limit of normal)
7. Unreliable social situation or inability to follow up
8. Contraindication to enoxaparin, warfarin and rivaroxaban
9. Atrial or ventricular dysrhythmia(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population is drawn from patients arriving in the Emergency Department who are then diagnosed with a lower risk pulmonary embolism (PESI score <86).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
90-day all-cause mortality, recurrent VTE, and Major Bleeding during outpatient treatment of Low-risk PE | 90 Days
  This is a composite outcome of the above.

SECONDARY OUTCOMES:
Reduction of medical costs due to outpatient treatment. | 90 Days
Level of patient satisfaction as measured by survey. | 90 Days Post study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bledsoe, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

REFERENCES:
- [Background] Aujesky D, Obrosky DS, Stone RA, Auble TE, Perrier A, Cornuz J, Roy PM, Fine MJ. Derivation and validation of a prognostic model for pulmonary embolism. Am J Respir Crit Care Med. 2005 Oct 15;172(8):1041-6. doi: 10.1164/rccm.200506-862OC. Epub 2005 Jul 14. PMID 16020800
- [Background] Aujesky D, Roy PM, Le Manach CP, Verschuren F, Meyer G, Obrosky DS, Stone RA, Cornuz J, Fine MJ. Validation of a model to predict adverse outcomes in patients with pulmonary embolism. Eur Heart J. 2006 Feb;27(4):476-81. doi: 10.1093/eurheartj/ehi588. Epub 2005 Oct 5. PMID 16207738
- [Background] Jimenez D, Yusen RD, Otero R, Uresandi F, Nauffal D, Laserna E, Conget F, Oribe M, Cabezudo MA, Diaz G. Prognostic models for selecting patients with acute pulmonary embolism for initial outpatient therapy. Chest. 2007 Jul;132(1):24-30. doi: 10.1378/chest.06-2921. PMID 17625081
- [Background] Squizzato A, Ageno W. The 8(th) American College of Chest Physicians Guidelines - a perspective on venous thromboembolism guidelines. Thromb Haemost. 2009 Jan;101(1):31-5. No abstract available. PMID 19132186
- [Background] Janjua M, Badshah A, Matta F, Danescu LG, Yaekoub AY, Stein PD. Treatment of acute pulmonary embolism as outpatients or following early discharge. A systematic review. Thromb Haemost. 2008 Nov;100(5):756-61. PMID 18989517
- [Background] Betriu A, Califf RM, Bosch X, Guerci A, Stebbins AL, Barbagelata NA, Aylward PE, Vahanian A, Van de Werf F, Topol EJ. Recurrent ischemia after thrombolysis: importance of associated clinical findings. GUSTO-I Investigators. Global Utilization of Streptokinase and t-PA [tissue-plasminogen activator] for Occluded Coronary Arteries. J Am Coll Cardiol. 1998 Jan;31(1):94-102. doi: 10.1016/s0735-1097(97)00428-2. PMID 9426024
- [Background] Koopman MM, Prandoni P, Piovella F, Ockelford PA, Brandjes DP, van der Meer J, Gallus AS, Simonneau G, Chesterman CH, Prins MH. Treatment of venous thrombosis with intravenous unfractionated heparin administered in the hospital as compared with subcutaneous low-molecular-weight heparin administered at home. The Tasman Study Group. N Engl J Med. 1996 Mar 14;334(11):682-7. doi: 10.1056/NEJM199603143341102. PMID 8594426
- [Background] Ageno W, Steidl L, Marchesi C, Dentali F, Mera V, Squizzato A, Crowther MA, Venco A. Selecting patients for home treatment of deep vein thrombosis: the problem of cancer. Haematologica. 2002 Mar;87(3):286-91. PMID 11869941
- [Background] Agnelli G, Verso M, Ageno W, Imberti D, Moia M, Palareti G, Rossi R, Pistelli R; MASTER investigators. The MASTER registry on venous thromboembolism: description of the study cohort. Thromb Res. 2008;121(5):605-10. doi: 10.1016/j.thromres.2007.06.009. Epub 2007 Aug 10. PMID 17692901
- [Background] Wells PS, Kovacs MJ, Bormanis J, Forgie MA, Goudie D, Morrow B, Kovacs J. Expanding eligibility for outpatient treatment of deep venous thrombosis and pulmonary embolism with low-molecular-weight heparin: a comparison of patient self-injection with homecare injection. Arch Intern Med. 1998 Sep 14;158(16):1809-12. doi: 10.1001/archinte.158.16.1809. PMID 9738611
- [Background] Wicki J, Perrier A, Perneger TV, Bounameaux H, Junod AF. Predicting adverse outcome in patients with acute pulmonary embolism: a risk score. Thromb Haemost. 2000 Oct;84(4):548-52. PMID 11057848
- [Background] Aujesky D, Obrosky DS, Stone RA, Auble TE, Perrier A, Cornuz J, Roy PM, Fine MJ. A prediction rule to identify low-risk patients with pulmonary embolism. Arch Intern Med. 2006 Jan 23;166(2):169-75. doi: 10.1001/archinte.166.2.169. PMID 16432084
- [Background] Brillman J, Mathers-Dunbar L, Graff L, Joseph T, Leikin JB, Schultz C, Severance HW Jr, Werne C. Management of observation units. American College of Emergency Physicians. Ann Emerg Med. 1995 Jun;25(6):823-30. doi: 10.1016/s0196-0644(95)70215-6. No abstract available. PMID 7755208
- [Background] Cross E, How S, Goodacre S. Development of acute chest pain services in the UK. Emerg Med J. 2007 Feb;24(2):100-2. doi: 10.1136/emj.2006.043224. PMID 17251613
- [Background] Daly S, Campbell DA, Cameron PA. Short-stay units and observation medicine: a systematic review. Med J Aust. 2003 Jun 2;178(11):559-63. doi: 10.5694/j.1326-5377.2003.tb05359.x. PMID 12765504
- [Background] Martinez E, Reilly BM, Evans AT, Roberts RR. The observation unit: a new interface between inpatient and outpatient care. Am J Med. 2001 Mar;110(4):274-7. doi: 10.1016/s0002-9343(00)00710-5. PMID 11239845
- [Background] Roberts R, Graff LG 4th. Economic issues in observation unit medicine. Emerg Med Clin North Am. 2001 Feb;19(1):19-33. doi: 10.1016/s0733-8627(05)70166-8. PMID 11214399
- [Background] Goodacre SW. Should we establish chest pain observation units in the UK? A systematic review and critical appraisal of the literature. J Accid Emerg Med. 2000 Jan;17(1):1-6. doi: 10.1136/emj.17.1.1. PMID 10658981
- [Background] Farkouh ME, Smars PA, Reeder GS, Zinsmeister AR, Evans RW, Meloy TD, Kopecky SL, Allen M, Allison TG, Gibbons RJ, Gabriel SE. A clinical trial of a chest-pain observation unit for patients with unstable angina. Chest Pain Evaluation in the Emergency Room (CHEER) Investigators. N Engl J Med. 1998 Dec 24;339(26):1882-8. doi: 10.1056/NEJM199812243392603. PMID 9862943
- [Background] Crenshaw LA, Lindsell CJ, Storrow AB, Lyons MS. An evaluation of emergency physician selection of observation unit patients. Am J Emerg Med. 2006 May;24(3):271-9. doi: 10.1016/j.ajem.2005.11.002. PMID 16635696
- [Background] Wilkinson K, Severance H. Identification of chest pain patients appropriate for an emergency department observation unit. Emerg Med Clin North Am. 2001 Feb;19(1):35-66. doi: 10.1016/s0733-8627(05)70167-x. PMID 11214403
- [Background] Dalen JE. Pulmonary embolism: what have we learned since Virchow? Natural history, pathophysiology, and diagnosis. Chest. 2002 Oct;122(4):1440-56. doi: 10.1378/chest.122.4.1440. No abstract available. PMID 12377877
- [Background] Goldhaber SZ, Elliott CG. Acute pulmonary embolism: part I: epidemiology, pathophysiology, and diagnosis. Circulation. 2003 Dec 2;108(22):2726-9. doi: 10.1161/01.CIR.0000097829.89204.0C. No abstract available. PMID 14656907
- [Derived] Bledsoe JR, Woller SC, Stevens SM, Aston V, Patten R, Allen T, Horne BD, Dong L, Lloyd J, Snow G, Madsen T, Elliott CG. Management of Low-Risk Pulmonary Embolism Patients Without Hospitalization: The Low-Risk Pulmonary Embolism Prospective Management Study. Chest. 2018 Aug;154(2):249-256. doi: 10.1016/j.chest.2018.01.035. Epub 2018 Feb 2. PMID 29410163